CLINICAL TRIAL: NCT00800566
Title: Phase I Study of Oral Clofarabine for the Treatment of Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: Oral Clofarabine in Chronic Lymphocytic Leukemia (CLL)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0905
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Chronic Lymphocytic Leukemia
Keywords: Clofarabine; Leukemia; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Clofarabine (Experimental)
  Interventions: Drug: Oral Clofarabine

INTERVENTIONS:
Drug: Oral Clofarabine — The starting dose will be 1 mg orally daily x 21 days every 4 weeks +/- 4 days.
  Other Names: Clolar®

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of clofarabine when given to patients with CLL. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Clofarabine is designed to interfere with the growth and development of cancer cells.

Screening Tests:

Before you can begin taking the study drug, you will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will also be asked about what drugs you are currently taking.
* You will be asked how well you are able to perform the normal activities of daily living (performance status evaluation).
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will also have a bone marrow aspirate and/or biopsy. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic and a small amount of bone marrow and bone is withdrawn through a large needle.
* Women who are able to have children must have a negative blood or urine pregnancy test. The blood would be drawn as part of the routine sample described above.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of clofarabine based on when you joined this study. Up to 7 dose levels of clofarabine will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of clofarabine is found.

The dose of clofarabine may be lowered or delayed to help reduce side effects.

Study Drug Administration:

On Days 1-21 of each 28-day study "cycle", you will take clofarabine by mouth once a day (in the morning) at about the same time everyday.

* You should take clofarabine on an empty stomach.
* You should try to fast (not eat anything or drink anything other than water) from midnight the night before each dose to 1 hour after taking clofarabine.
* Clofarabine should be taken with 4 ounces (1/2 a cup) of water.
* You should not drink coffee and other caffeinated liquids before and for 1 hour after taking the study drug.
* If you vomit more than 15 minutes after you take the drug, you should not replace or make up the drug. If you vomit less then 15 minutes after taking the drug, you should retake the dose. If you vomit again within 15 minutes after retaking the dose, you should not take the drug again that day and make a note of it in the diary.

Study Visits:

* On Day 1 of every cycle, the following tests and procedures will be performed:
* You will have a physical exam, including measurement of your weight and vital signs.
* You will have a performance status evaluation.
* You will be asked if you have experienced any intolerable side effects and how you are feeling.

Once a week of Cycle 1, you will have a physical exam.

Once a week of every cycle, blood (about 1-2 teaspoons) will be drawn for routine tests (blood counts with platelets). Your blood will be drawn more often if the doctor feels it is necessary.

After Cycles 3 and 6, you will have a bone marrow aspiration and/or biopsy to check the status of the disease.

If you go off study before Cycle 3 and the doctor thinks it is necessary, the bone marrow aspiration and/or biopsy may be taken when you go off study.

If you have completed all 6 cycles of the study drug, every 6 months (+/- 2 months), you will have a physical exam and blood (about 1-2 teaspoons) will be drawn to check on the status of the disease and your overall health. The study doctor will tell you any other tests that may be needed.

Length of Study You will be on the study drug for up to 6 cycles (about 6 months). You will be taken off study early if the disease gets worse or you experience any intolerable side effects.

Additional Information:

You will need to stay in Houston for Cycle 1 (28 days). After that, you may return to your home but you will still have to return to Houston before each cycle unless you choose to have check-up visits and blood tests with your local doctor.

This is an investigational study. Clofarabine is FDA approved and commercially available when given by vein to pediatric patients for the treatment of acute lymphoblastic leukemia (ALL) that has come back or not responded to other treatments. The use of clofarabine by mouth is not FDA approved. At this time, oral clofarabine is only being used in research.

Up to 36 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lymphocytic leukemia (CLL), CLL/PLL (as defined by FAB [French-American-British Classification]), small lymphocytic lymphoma (SLL) and prolymphocytic leukemia (PLL) who have relapsed from or are refractory to at least one fludarabine-based regimen and no greater than 2 regimens.
* Absolute neutrophil count (ANC) >= 1 x 109/L and platelet count >= 50 x 109/L.
* Adequate organ function as indicated by the following laboratory values: serum creatinine </= 1 mg/dL; if serum creatinine > 1 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 ml/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation; serum bilirubin </= 1.5 mg/dL x ULN; aspartate transaminase (AST)or alanine transaminase (ALT) </= 2.5 x ULN; alkaline phosphatase </= 2.5 x ULN.
* ECOG performance status <= 2.
* Age >/= 18 years.

Exclusion Criteria:

* Patients with NYHA >/= grade 3 heart disease as assessed by history and/or physical examination.
* Pregnant or breastfeeding women or patients who are unwilling or unable to practice adequate contraception. Positive pregnancy test for women of child bearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization).
* Chemotherapy within 4 weeks of starting therapy, or concurrent anticancer therapy (chemotherapy, radiotherapy, or biologic therapy).
* Other malignancy within 3 years except in situ carcinoma.
* Unwilling or unable to provide informed consent.
* Known hypersensitivity to nucleoside analogues.
* Any other significant medical condition that compromises safety, compliance or study conduct, including but not limited to uncontrolled hypertension, unstable angina, myocardial infarction within 6 months, ventricular arrhythmia, active infection, and known hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and Dose limiting toxicities (DLT) | October 2009

SECONDARY OUTCOMES:
To investigate the plasma clofarabine and cellular clofarabine triphosphate pharmacology profile in CLL. | October 2010

CONTACTS AND LOCATIONS:
Overall Officials: Stefan F. Faderl, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's Website — http://mdanderson.org